CLINICAL TRIAL: NCT00337142
Title: Follow up Glucose Levels Among Infants of Diabetic Mothers
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Ayala Maayan, Sheba Medical Center
Other Study IDs: SHEBA-06-4266-AM-CTIL
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Newborn; Full Term; Diabetic Mother
Keywords: gestational diabetes; newborn; hypoglycemia
MeSH Terms: conditions — Diabetes, Gestational; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Infants to diabetic mothers (IDM) are at risk for developing hypoglycemia after birth. Glucose level follow ups are recommended to each IDM. However, there are no recommendations as to how long this follow up should be performed for, nor are there "safe" glucose levels that allow stopping glucose monitoring.

The aim of the study is to retrospectively follow up glucose levels among IDMs in order to find risk factors for developing hypoglycemia and determine time and glucose levels that would permit monitoring cessation.

DETAILED DESCRIPTION:
A retrospective study of 250-300 IDMs, born in a single large medical center. Data will be collected as follows: Gestational age, birth weight, sex, delivery mode, type of maternal diabetes, other maternal diseases, feeding mode. Glucose levels as were recorded according to newborn protocol (1,2,4,6 hours after delivery, and then every 8 hours for total of 48 hours). Data of hypoglycemia treatment, if given, will be collected.

Later we will statistically try to determine the risk factors for developing hypoglycemia and the "safe" time and glucose levels to stop monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Full-term infants, diabetic mothers, Singleton

Exclusion Criteria:

* Preterm infants, multiple pregnancy, congenital malformations, clinically ill at birth.

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Maayan, MD, Principal Investigator — Sheba Medical Center